CLINICAL TRIAL: NCT03641066
Title: The Effect of Progressing Ankle Brace Restriction on Walking and Running Gait Characteristics in Healthy Individuals
Brief Title: Progressing Ankle Brace Restriction on Walking and Running Gait Characteristics in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sport and Spine Rehab Clinical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AnkleBrace Running
Record Dates: First submitted 2018-07-02; First posted 2018-08-21 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Ankle Sprains
Keywords: ankle; biomechanics
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ankle Brace (Experimental): Each participant will complete a baseline analysis of 1 minute of walking and 2 minutes of running, repeated 4 more times wearing 4 different braces. The analysis will be completed on the Walker View Treadmill, which used 3D camera technology to capture lower body kinematics. The treadmill also has load cells built in to capture gait characteristics
  Interventions: Device: Ankle Brace

INTERVENTIONS:
Device: Ankle Brace — Each participant will complete the 1 minute walking and 2 minute running under 5 conditions [1] un-braced, [2] Active Ankle 329 Ankle Sleeve, [3] AS1Pro (a lace-up brace), [4] Eclipse 1 (single-upright brace), and [5] Eclipse 2 (double upright brace)

SUMMARY:
A convenience sample of 20 participants, 18 years or older healthy individuals were recruited. Participants were excluded if they report being pregnant or being treated for a musculoskeletal injury. After explanation of the study and consent were obtained, each participant completed background information and the Cumberland Ankle Instability Tool (CAIT). Participants began by completing a 1 minute, 3mph walking gait assessment while unbraced, followed by a 2-minute, 6mph unbraced running assessment. Following the unbraced condition participants were randomly assigned into 1 of 4 conditions: [1] Active Ankle 329 Ankle Sleeve, [2] AS1Pro, [3] Eclipse 1, or [4] Eclipse 2. Participants placed an assigned brace on each ankle and then repeated the walking gait and running assessments. After this test the participants filled out a 10-item satisfaction questionnaire, and then were randomly assigned a second brace. The protocol was repeated until they have completed the walking, running, and satisfaction survey in all 4 brace conditions.

DETAILED DESCRIPTION:
A convenience sample of 20 participants, 18 years or older healthy individuals were recruited. Participants were excluded if they report being pregnant or being treated for a musculoskeletal injury. After explanation of the study and consent were obtained, each participant completed background information and the Cumberland Ankle Instability Tool (CAIT). Participants began by completing a 1 minute, 3mph walking gait assessment while unbraced, followed by a 2-minute, 6mph unbraced running assessment. Following the unbraced condition participants were randomly assigned into 1 of 4 conditions: [1] Active Ankle 329 Ankle Sleeve, [2] AS1Pro, [3] Eclipse 1, or [4] Eclipse 2. Participants placed an assigned brace on each ankle and then repeated the walking gait and running assessments. After this test the participants filled out a 10-item satisfaction questionnaire, and then were randomly assigned a second brace. The protocol was repeated until they have completed the walking, running, and satisfaction survey in all 4 brace conditions.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals who are able to run for 10 minutes total

Exclusion Criteria:

* pregnancy, lower body injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Ankle Dorsiflexion/Plantarflexion Range of Motion | Ankle Dorsiflexion/Plantarflexion Range of Motion will be measured for the last 30 seconds of the 1 minute walk, and the last 30 seconds of the 2 minute run. It will be measured during each of the 5 conditions.
  Ankle Dorsiflexion/Plantarflexion Range of Motion will be measured using the Woodway Walker View Treadmill which utilizes a 3D camera
Change in Ankle Inversion/Eversion Range of Motion | Ankle Inversion/Eversion Range of Motion will be measured for the last 30 seconds of the 1 minute walk, and the last 30 seconds of the 2 minute run. It will be measured during each of the 5 conditions.
  Ankle Inversion/Eversion Range of Motion will be measured using the Woodway Walker View Treadmill which utilizes a 3D camera
Change in Knee Flexion Range of Motion | Knee Flexion Range of Motion will be measured for the last 30 seconds of the 1 minute walk, and the last 30 seconds of the 2 minute run. It will be measured during each of the 5 conditions.
  Knee Flexion Range of Motion will be measured using the Woodway Walker View Treadmill which utilizes a 3D camera
Change in Step Length | Step Length will be measured for the last 30 seconds of the 1 minute walk, and the last 30 seconds of the 2 minute run. It will be measured during each of the 5 conditions.
  Step Length will be measured using the Woodway Walker View Treadmill which utilizes load cells within the treadmill belt

CONTACTS AND LOCATIONS:
Locations (1):
- Sport & Spine Rehab, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No